CLINICAL TRIAL: NCT05308459
Title: Data Driven Health Promotion at Vocational Education and Training Schools (The Data Health VET Study)
Brief Title: Data Health VET - Data-driven Health Promotion at Vocational Education and Training Schools
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Steno Diabetes Center Sjaelland (Other Government); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Charlotte Demant Klinker, Senior researcher, Steno Diabetes Center Copenhagen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Data Health VET
Record Dates: First submitted 2022-03-08; First posted 2022-04-04 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Food Habits; Physical Inactivity; Smoking Behaviors; Drug Use; Alcohol Consumption; Wellbeing
Keywords: Vocational school; Health behavior; Organizational Readiness; Health promotion
MeSH Terms: conditions — Feeding Behavior; Sedentary Behavior; Smoking; Alcohol Drinking; Health Behavior

STUDY DESIGN:
Intervention Model Description: A non-randomized clustered stepped-wedge design with two steps will be applied. Four VET schools (one from each of the four main educations tracks) are selected to early start (January 2022) and four to late start - also one from each of the four main educational tracks (6 months later). This design allows the intervention to be rolled out sequential, allowing us to control for differences between study sites (vertical control) and secular trends (horizontal control) during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step 1: Allocated to start the Data Health VET intervention phase January 2022 (Experimental): Participants receive the Data Health VET intervention in all its steps starting in January 2022
  Interventions: Behavioral: Data-driven health promotion at Vocational Education and Training schools (Data Health VET)
- Step 2: Allocated to start the Data Health VET intervention phase August, 2022 (Experimental): Participants receive the Data Health VET intervention in all its steps starting in August 2022
  Interventions: Behavioral: Data-driven health promotion at Vocational Education and Training schools (Data Health VET)

INTERVENTIONS:
Behavioral: Data-driven health promotion at Vocational Education and Training schools (Data Health VET) — The intervention consists of the following steps:
  1. A local health profile is conducted among all students
  2. Results are shortly hereafter presented and discussed with all student and staff, and the school decide what health problem they will work with during the next year
  3. A participatory group model process based on a dynamic systems approach is conducted to develop sustainable and system changing activities to address the chosen health problem
  4. The activities are implemented
  5. A new health profile is conducted to a) evaluate the effects of the implemented activities and to b) determine if a new health problem warrant focus and new activities are needed (the process repeats itself).

SUMMARY:
The purpose of this study is to investigate the effectiveness of a data driven and dynamic systems approach at Danish Vocational schools to promote student health behavior and wellbeing and school organizational readiness.

DETAILED DESCRIPTION:
Background:

Recent evidence shows that vocational education and training (VET) school students exhibits significant risk behaviors in terms of poor diet, frequent smoking, low levels of physical activity and poor mental health.

Health behavior constitutes a complex problem that is influenced by underlying, dynamic mechanisms and determinants at multiple levels. A system perspective is an evidence-based approach that has the potential to address and initiate sustainable changes to complex health problems, but studies are needed to translate, test, and adapt such evidence-based methods to the VET school setting.

Objective:

Data driven Health promotion at Vocational Education and Training schools (the Data Health VET study) aims to develop a sustainable model to promote health and wellbeing among vocational school students. The objective of this study is to investigate the effectiveness of the model.

Design:

A non-randomized clustered stepped-wedge design will be applied. Eight intervention schools will be included in two steps:

Step 1: early starters (January 2022) Step 2: late starters (August 2022).

Intervention:

The intervention consists of the following steps:

1. A local health profile is conducted among all students
2. Results are shortly hereafter presented and discussed with all student and staff, and the school decide what health problem they will work with during the next year
3. A participatory group model process based on a dynamic systems approach is conducted to develop sustainable and system changing activities to address the chosen health problem
4. The activities are implemented
5. A new health profile is conducted to a) evaluate the effects of the implemented activities and to b) determine if a new health problem warrant focus and new activities are needed (the process repeats itself).

Participants:

The eight intervention schools are located in the capital region of Denmark and Region Zealand and have been recruited so each region participates with one school from each of four, main vocational educational tracks: 1) technical (e.g. electrician), 2) business (e.g. office assistant), 3) agriculture and food service (e.g. farmer or chef) and 4) social and health service (e.g. health service assistant). Across the eight intervention schools the target population is estimated to be at student level n=1800, staff members and mangers: n≈160, other involved local partners (n≈80). All are eligible for both intervention and evaluation.

Study measures:

The study investigates 1) changes in student's health behaviour and wellbeing and 2) changes in organizational motivation and capacity to work with and implement health promotion initiatives. The primary and secondary student outcome measure for each cluster depends on the chosen health promotion theme. Moreover, the study explores if the intervention influences different student health promotion outcomes (e.g. health literacy, motivation, knowledge).

Data Health VET will provide solid evidence of the effects of the Data Health VET model, which is needed in practice to inform the scale-up of the model to other VET schools or settings. The study is conducted in partnership between the applying institutions and the participating schools and municipalities through all phases.

ELIGIBILITY:
Inclusion Criteria:

* All employees at the participating schools
* All students who are at the school at the time for data collection
* Participants who have provided written informed consent.

Exclusion Criteria:

* Schools which do not develop and implement any activities that aim to promote health among the students will be excluded from the analysis on student level but will be included in the analysis on organizational level.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1370 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Wellbeing during schooltime (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured by asking participants how they feel about school at present
Physical activity level during schooltime (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured using the Saltin-Grimby Physical Activity Level Scale (SGPALS) adapted to the school setting
Food intake during schooltime (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured using an adapted version of dietary behavior used in the large national and international Health Behavior in School-aged Children (HBSC) survey. Participants will be asked about their frequency in which they consumed various food during school time on a normal school week
Tobacco use during schooltime (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured by asking the participants if they smoke cigarettes, e-cigarettes or uses snuff or other tobacco products during schooltime
Alcohol consumption during schooltime (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured by asking the participants if they consume alcohol during schooltime
Marihuana and drug use during schooltime (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured by asking the participants if they use the products during schooltime
Organizational Readiness (organizational outcome) | The questionnaire will be distributed among the school staff at baseline, T1 (6 months), T2 (12 months) and T3 (24 months).
  Changes in the schools Organizational Readiness (OR) is measured using a questionnaire instrument measuring 1) Organizational motivation, 2) General capacity and 3) Health Promotion Capacity as proposed in Scaccia et al. 2015's organizational readiness theory. The three domains are predominantly measured using validated scales with some adjustments and additions to comply with the study and setting.

SECONDARY OUTCOMES:
Wellbeing (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured using WHO-5 questionnaire
Physical activity (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured using the SGPALS
Food intake (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured using an adapted version of dietary behavior used in the HBSC survey. Participants will be asked about their frequency in which they consumed various food on a normal week
Tobacco use (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured by asking the participants if they smoke cigarettes, e-cigarettes or uses snuff or other tobacco products
Alcohol consumption (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in Binge drinking will be measured by asking participants how often they have been drinking 5 or more drinks on the same occasion in the past 30 days
Marihuana and drug use(student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes will be measured by asking the participants how often they have used the products the past 30 days

OTHER OUTCOMES:
Health Literacy (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in students health Literacy (HL) is measures using the Health Literacy for School-Aged Children (HLSAC) questionnaire (10 items).
Knowledge relevant to the problem of interest (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in knowledge relevant to the problem of interest (wellbeing, physical activity, healthy food intake, smoking, alcohol) will be measured by 5 self-developed items, specified from the knowledge question from HLSAC.
Behavioral intentions (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in behavioral intentions will be measured using 5 items from The Danish National Health Survey.
Motivation (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in motivation relevant to the problem of interest (physical activity, healthy food intake, smoking, alcohol) will be measured by 4 items from The Danish National Health Survey.
Social connectedness (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in social connectedness will be measured by tree items used in the HBSC survey.
Self-empowerment (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in self-empowerment will be measured using the Actively managing my health domain from Health Literacy Questionnaire (HLQ) (5 items)
Self-confidence (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in self-confidence (self-efficacy and self-esteem) will be measured with two items used in the HBSC survey.
Student autonomy (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in student autonomy will be measured by two items adapted from the HBSC survey.
Social relationships (student outcome) | Baseline, T1 (12 months), T2 (18 months) and T3 (24 months)
  Changes in social relationships will be measured by two items from The Danish National Health Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte D Klinker, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Herlev
  - Steno Diabetes Center Zealand, Holbæk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinze C, Hartmeyer RD, Sidenius A, Ringgaard LW, Bjerregaard AL, Krolner RF, Allender S, Bauman A, Klinker CD. Developing and Evaluating a Data-Driven and Systems Approach to Health Promotion Among Vocational Students: Protocol for the Data Health Study. JMIR Res Protoc. 2024 Feb 6;13:e52571. doi: 10.2196/52571. PMID 38319698